CLINICAL TRIAL: NCT02588547
Title: Prophylactic Granisetron for the Prevention of Spinal Induced Shivering During Cesarean Section: a Prospective Double Blind Dose Ranging Clinical Study
Brief Title: Prevention of Spinal Induced Shivering During CS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM102015
Record Dates: First submitted 2015-10-24; First posted 2015-10-28 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Spinal Induced Shivering
Keywords: Shivering; Granisetron; Spinal; Cesarean section
MeSH Terms: interventions — Granisetron; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Granisetron 1 (Active Comparator): Intravenous granisetron 1 mg
  Interventions: Drug: Granisetron
- Granisetron 0.7 (Active Comparator): Intravenous granisetron 0.7 mg
  Interventions: Drug: Granisetron
- Placebo (Placebo Comparator): intravenous 0.9% Sodium chloride (2 ml)
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Granisetron — IV granisetron 1 mg before spinal anethesia
  Other Names: Kytril ampule 3mg/3ml IV (Roche)
  Arms: Granisetron 1
Drug: Granisetron — IV granisetron 0.7 mg before spinal anethesia
  Other Names: Kytril ampule 3mg/3ml IV (Roche)
  Arms: Granisetron 0.7
Drug: Sodium chloride — IV 2 ml 0.9 sodium chloride before spinal anethesia
  Other Names: 0.9 Sodium chloride
  Arms: Placebo

SUMMARY:
This study compares the efficacy of two different doses of intravenous (IV) granisetron on the prevention of postspinal shivering during cesarean section, in comparison with placebo.

DETAILED DESCRIPTION:
The study will includes four groups as follows:

1. Granisetron1 group: women will receive 1mg IV granisetron
2. Granisetron 0.7 group: women will receive 0.7 mg IV granisetron and
3. Control group: women will receive 2 ml of 0.9% sodium chloride. Throughout the study period,shivering scores, core temperature, sensory level and motor block will be recorded, heart rate will be measured continuously using an electrocardiogram; blood pressure will be determined. If heart rate decreases by more than 20% of the baseline atropin will be received and if blood pressure decreases 20% of the baseline ephedrine will be received.

Also, Apgar score at one minute and five minutes will be recorded. At the end patient satisfaction will be assessed using Verbal Numeric Scoring system Side effects (bradycardia, hypotension, hypothermia, nausea and vomiting, pruritus etc ) will be recorded perioperatively in the operating room and postanesthetic care unit.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at term,
* ASA status I or II (American Society of Anesthesiologists) physical status class I-II,
* low-risk cesarean section,
* Scheduled for the spinal anesthesia

Exclusion Criteria:

* Pregnant women in labor
* Patients who have the body temperature over 37.3 or less than 37 celsius degree
* Known allergies to the study drugs
* Contraindication to spinal anesthesia

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 212 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
shivering score | 180 min (immediately before the block till 180 min after the block)

SECONDARY OUTCOMES:
non invasive blood pressure | 90 min (immediately before the block till 90 min after the block)
heart rate | 90 min (immediately before the block till 90 min after the block)
core temperature | 90 min (immediately before the block till 90 min after the block)

CONTACTS AND LOCATIONS:
Overall Officials: Seham M Moeen, MD, Principal Investigator — Assiut Univerisity
Locations (1):
- Seham Mohamed Moeen Ibrahim, Asyut, Egypt

REFERENCES:
- [Derived] Abdel-Ghaffar HS, Moeen SM. Prophylactic granisetron for post-spinal anesthesia shivering in cesarean section: A randomized controlled clinical study. Acta Anaesthesiol Scand. 2019 Mar;63(3):381-388. doi: 10.1111/aas.13084. Epub 2018 Feb 8. PMID 29424008